CLINICAL TRIAL: NCT02743416
Title: Systematic NT-proBNP and ECG Screening for Atrial Fibrillation Among 75 Year Old Subjects in the Region of Stockholm, Sweden - STROKESTOP II
Acronym: STROKESTOP II
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Principal Investigator, Professor Mårten Rosenqvist, Professor, Karolinska University Hospital
Other Study IDs: STROKESTOP II
Record Dates: First submitted 2016-03-16; First posted 2016-04-19 (Estimated); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: Screening; Stroke prevention; Cost effectiveness
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — venous blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ECG screening: Will be screened for AF using only one-stop protocol
  Interventions: Other: ECG screening (Zenicor-ECG) for atrial fibrillation
- Control group: as per regular standard as of today

INTERVENTIONS:
Other: ECG screening (Zenicor-ECG) for atrial fibrillation — Determination of the biomarker NT-proBNP together with single-lead ECG screening for silent atrial fibrillation.
  Groups: ECG screening

SUMMARY:
STROKESTOP II will study if the biomarker NT-proBNP together with single-lead ECG can be used as a primary population screening tool for silent atrial fibrillation, and builds on previous results from the STROKESTOP study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals born 1940 and 1941 residing in Stockholm at the time of inclusion

Exclusion Criteria:

* Not fulfilling the inclusion criteria

Ages: 75 Years to 76 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Individuals aged 75/76 residing in Stockholm will be identified using their 10-digit personal identification number. All identified subjects will be randomized in a 1:1 fashion to be invited to screening for AF or to serve as a control group.
  Participants with a prior diagnosis of AF will be asked if they are on treatment with anticoagulants. If they are not, a referral to cardiologist will be made to ensure appropriate treatment.
  Individuals without known AF will have blood samples drawn and analysed with regard to NT-proBNP using point of care analysis.
  All individuals with NT-proBNP> 125 ng/L and without known AF will be taught to undergo intermittent ECG recordings twice daily for two weeks (High-risk Group). Individuals with a NT-proBNP<125 ng/L will do one initial 1-lead ECG, and if normal not undergo further ECG screening (low-risk Group).
Sampling Method: Probability Sample
Enrollment: 6868 (Actual)
Dates: Start 2016-04; Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of stroke or systemic embolism in the control group vs the intervention group | Five years
  Endpoints collected from the Swedish patient registry will be compared between the groups
Incidence of stroke or systemic embolism in the control group vs the low-risk group (with NT-proBNP<125 ng/L and normal index 1-lead ECG). | Five years
  Endpoints collected from the Swedish patient registry will be compared between the groups

SECONDARY OUTCOMES:
Incidence of major bleeding, ischaemic stroke, systemic embolism and death in the control group vs the intervention group | Five years
  Endpoints collected from the Swedish patient registry will be compared between the groups
Number of subjects with new discovered AF using intermittent ECG-recordings in the high risk Group with NT-proBNP>125 ng/L. | Two years
  All individuals with NT-proBNP>125ng/L will undergo intermittent ECG recordings at least twice daily for two weeks.
To assess screening uptake with regards to socio-demographic factors and to study if we can improve uptake in the screening programme by decentralizing the recruitment procedure. | Two years
  Participants and non-participants will be compared using socioeconomic data provided by statistics sweden
Cost per gained quality-adjusted life-year (QALY) and cost per avoided stroke of the STROKESTOP II screening program. | Five years
  With the same statistical methods used in STROKESTOP I, the number of fewer years with undetected AF will be calculated as well as the number of avoided strokes, the number of life-years and the number of quality-adjusted life years (QALYs) per 1000 screened patients. The result will be reported as the incremental cost per gained QALY and per avoided stroke.
Plasma and serum biomarkers and their relation to incidence of new AF and short episodes of AF (micro-AF) | Five years
  serum and plasma biomarkers within coagulation, inflammation, cardiomyocyte stress, atrial fibrosis, electrical remodelling, prothrombotic state and altered haemodynamics will be analysed with immunoassays, in order to identify the best discriminator for silent AF on population level. https://www.olink.com/products/cvd-iii-panel/
To assess the incidence of heart failure in patients with NT-proBNP>125ng/L | Five years
  To assess the value of structured follow-up with echocardiography in participants without known heart failure, but with increased NT-proBNP as a method to diagnose heart failure with reduced and preserved ejection fraction; and to assess whether in patients with NT-proBNP > 125 pg/mL, a higher cut-off can be used to predict HF on echocardiography, and thus be used to triage asymptomatic patients to echocardiography.
To study atrial function in patients with and without silent atrial fibrillation | Five years
  In a subset of participants with and without atrial fibrillation, advanced atrial echocardiography will be performed
To study the correlation between symptoms and newly discovered AF | Four years
  Participants are asked if they have had symptoms of palpitations before screening visit
To study the diagnostic performance of pulse-palpation in AF screening as compared to one-lead ECG | Four years
  pulse palpation will be performed in all participants and then a single-lead ECG will be registered
To study the association of very short episodes of AF (micro-AF, episodes lasting shorter than 30 seconds) and incident AF | Two years
  Individuals with micro-AF, defined as at least five supraventricular ectopics in a row but lasting shorter than 30 seconds at any time during intermittent screening will be compared to participants without micro-AF with regard to incident AF during screening.
To compare different ECG modalities for AF screening | Two years
  A subset of participants will perform both single-lead, handheld, intermittent ECG (Zenicor) and continuous event loop ECG recordings (Novacor R-test 4) and AF yield (defined as at least one episode of AF with a duration of 30 seconds) will be compared between the methods. Tolerability to both methods will be measured qualitatively with a questionnaire.
Incidence of undiagnosed hypertension in participants | four years
  Blood pressure will be measured and participants with elevated blood pressure but no previous diagnosis of hypertension will be referred for further evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Mårten Rosenqvist, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Trial Alliance, KTA Prim, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kemp Gudmundsdottir K, Svennberg E, Friberg L, Hygrell T, Frykman V, Al-Khalili F, Hijazi Z, Rosenqvist M, Engdahl J. Randomized Invitation to Systematic NT-proBNP and ECG Screening in 75-Year-Olds to Detect Atrial Fibrillation: STROKESTOP II. Circulation. 2024 Dec 3;150(23):1837-1846. doi: 10.1161/CIRCULATIONAHA.124.071176. Epub 2024 Sep 1. PMID 39217615
- [Derived] Fredriksson T, Gudmundsdottir KK, Frykman V, Friberg L, Al-Khalili F, Engdahl J, Svennberg E. Brief episodes of rapid irregular atrial activity (micro-AF) are a risk marker for atrial fibrillation: a prospective cohort study. BMC Cardiovasc Disord. 2020 Apr 10;20(1):167. doi: 10.1186/s12872-020-01453-w. PMID 32276611